CLINICAL TRIAL: NCT03061006
Title: Impact of Anticoagulation Therapy on the Cognitive Decline and Dementia in Patients With Non-Valvular Atrial Fibrillation (CAF Trial)
Brief Title: Impact of Anticoagulation Therapy on the Cognitive Decline and Dementia in Patients With Non-Valvular Atrial Fibrillation
Acronym: CAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1050164
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Dementia; Cognition Disorders; Cerebral Ischemic Events
MeSH Terms: conditions — Dementia; Cognition Disorders | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabigatran Etexilate (Experimental): 150 mg BID (CrCL > 30 mL/min) or 75 mg BID (CrCL 15-30 mL/min)
  Interventions: Drug: Dabigatran Etexilate
- Warfarin (Active Comparator): Dose-adjusted warfarin (INR: 2.0-3.0)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran Etexilate — 150 mg BID (CrCL > 30 mL/min) or 75 mg BID (CrCL > 15 to 30 mL/min); Assessment of kidney function every 6 months.
  Other Names: Pradaxa
  Arms: Dabigatran Etexilate
Drug: Warfarin — Dose-adjusted (INR 2.0 - 3.0); Standard warfarin follow-up and education based upon system criteria.
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
Patients will be screened at Intermountain Medical Center and at Intermountain-affiliated anticoagulation clinics in the Salt Lake City region. Patients with non-valvular atrial fibrillation will be considered for study. After written informed consent is obtained, subjects who meet eligibility criteria will be randomized 1:1 to 2 treatment arms: Group 1: Dabigatran etexilate (150 mg BID if CrCL > 30 mL/min, or 75 mg BID if CrCL > 15 to 30 mL/min or per USPI; and Group 2: Warfarin (Dose-adjusted (INR 2.0 - 3.0). Assessment of kidney function every 6 months will be done for Group 1. Standard warfarin follow-up and education, based upon system criteria, will be done for Group 2. All subjects will be followed for 24 months, and will be assessed at 1-week, then 3-, 6-, 12-, 18- and 24-months post-anticoagulation visits as well as other visits deem necessary for clinical care. All subjects will undergo protocol-specified laboratory tests and will complete 6 standard, validated questionnaires at each follow-up visit following the week 1 visit, except at the 3-month visit when only one questionnaire will be administered. To determine brain volume and characteristic changes representative of micro-bleeding, the first 10 subjects in each treatment group who are willing and able to undergo the procedure will participate in a MRI sub-study. The cranial MRI will be done at baseline and at 24-months post-anticoagulation on this sub-group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >65 years of age.
2. Non-valvular atrial fibrillation documented by electrocardiogram, ambulatory event monitor, or telemetry within 12 months of enrollment.
3. Moderate risk of thromboembolism based upon a CHADS score or CHADS2 Vasc score of ≥2.
4. Ability to complete a mini-mental status evaluation.
5. Ability to independently comprehend and complete a quality of life and dementia questionnaires.
6. Ability to provide informed consent for study participation.
7. Willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

1. Inability to take an anticoagulant due to known or perceived bleeding risk.
2. Known coagulopathy that may impact the choice, duration, efficacy and safety of anticoagulation therapy.
3. Atrial Fibrillation in the setting of valvular heart disease. Valvular heart disease defined as any surgical valve, mitral stenosis, or moderate-severe valvular heart disease.
4. Severe renal dysfunction, defined as a creatinine clearance rate <15 mL/min (documented within the last 3 months).
5. History of any form of dementia.
6. A life expectancy less than 24 months.
7. Inability to comply with the follow-up schedule.
8. Current participation in a clinical investigation that includes an active pharmacologic treatment arm.
9. An upper age limit not to be used if participation inclusion criteria are met.
10. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.
11. Other conditions that in the opinion of the Principal Investigator(s) may increase risk to the subject and/or compromise the quality of the clinical trial.
12. Concurrent pharmacologic treatment that is required to treat a condition long-term in which concurrent use of dabigatran etexilate is contraindicated.
13. Treatment with any anticoagulant drug for stroke prevention for more than 30 days.

    * Aspirin and P2Y12 inhibitors (e.g. clopidogrel (Plavix), or prasugrel (Effient)) are not considered anticoagulant drugs.
    * If the subject has received any anticoagulant drug for stroke prevention for less than 30 days, the Principal Investigator(s) or a Co-Investigator will decide whether or not the subject is eligible for this study
14. The Principal Investigator(s) determine(s) that the subject is not eligible for participation in this research study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Incident dementia determined by a formal diagnosis of dementia by a neurologist | 24 months
  Incident dementia will be determined by a formal diagnosis of dementia by a neurologist
Moderate decline in cognitive function based on results of the Alzheimer's Disease Assessment Scale and the Disability Assessment for Dementia. | 24 months
  Determined by measuring the change from baseline to study conclusion on the 11-item cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-cog11, with scores ranging from 0 to 70, and higher scores indicating greater impairment) and the Disability Assessment for Dementia (DAD, with scores ranging from 0 to 100, and higher scores indicating less impairment). An increase in ADAS-cog11 of >30% is considered significant for moderate cognitive decline. In subjects that score <50% on the DAD, there is a direct correlation with global deterioration scales and scores. Subjects with a 30% decrease in DAD score or those with a score <50% will be considered to have moderate cognitive decline. These scores will be aggregated and if a patient meets either one of the cognitive decline definitions they will be deemed positive for cognitive impairment.

SECONDARY OUTCOMES:
Stroke or Transient ischemic attack (TIA), intracranial bleed | 24 months
Changes from baseline scores on the mini-mental status evaluation and the Hachinski Ischemic Scale. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States

REFERENCES:
- [Derived] Kwan J, Hafdi M, Chiang LLW, Myint PK, Wong LS, Quinn TJ. Antithrombotic therapy to prevent cognitive decline in people with small vessel disease on neuroimaging but without dementia. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD012269. doi: 10.1002/14651858.CD012269.pub2. PMID 35833913